CLINICAL TRIAL: NCT04031339
Title: Multicenter, Prospective, Observational Study of Clinical Outcomes of Thyroid Cancer
Brief Title: Study of Clinical Outcomes of Thyroid Cancer
Acronym: ITCO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Italian Thyroid Cancer Observatory (ITCO) Foundation (Unknown); Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Sebastiano Filetti, Full Professor of Internal Medicine, University of Roma La Sapienza
Other Study IDs: 3366
Record Dates: First submitted 2019-06-25; First posted 2019-07-24 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Thyroid Neoplasms
Keywords: papillary thyroid cancer; follicular thyroid cancer; poorly differentiated thyroid cancer; anaplastic thyroid cancer; medullary thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary; Adenocarcinoma, Follicular; Thyroid Carcinoma, Anaplastic; Carcinoma, Medullary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with thyroid cancer: Patients with histologically-confirmed diagnoses of papillary, follicular, Hürthle, poorly differentiated, anaplastic, or medullary thyroid cancer
  Interventions: Procedure: Standard treatment

INTERVENTIONS:
Procedure: Standard treatment — e.g., surgery, radioiodine therapy, systemic treatments (multikinase inhibitors), surveillance

SUMMARY:
The Italian Thyroid Cancer Observatory (ITCO) repository was established to collect data on thyroid cancer management in a prospective and consecutive series of newly-diagnosed patients, enrolled in centers uniformly distributed across the nation.

DETAILED DESCRIPTION:
Little information is available on current practices in the treatment of thyroid cancer: a web-based thyroid cancer database was created to collect real-life data. The participants' network include tertiary referral centers operating at the national level, as well as smaller hospital-based units with local or regional recruitment areas.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed thyroid cancer
* clinical follow-up including serum thyroglobulin (Tg) assays, circulating Tg antibodies, and high-resolution gray-scale and color Doppler US of the thyroid bed and cervical lymph node compartments. Additional imaging studies and/or fine-needle aspiration biopsy for cytology are ordered at the examiner's discretion in accordance with evidence-based guidelines
* entire follow-up at a participating clinical center.

Exclusion Criteria:

* patients referred to the recruiting centers ≥12 months from the primary treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients prospectively and consecutively diagnosed with histologically-confirmed papillary, follicular, Hürthle, poorly differentiated, anaplastic, or medullary thyroid cancer.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Disease persistence or recurrence | Up to 10 years from the primary treatment
  Composite event of disease persistence or recurrence during clinical follow-up, detected by any of the available imaging tools (neck sonography, computed tomography [CT], magnetic resonance imaging [MRI], or positron emission tomography [PET])

SECONDARY OUTCOMES:
Disease persistence after 12-18 months from the primary treatment | 12-18 months from the primary treatment
  Rate of disease persistence after 12-18 months from the primary treatment, detected by any of the available imaging tools (neck sonography, radioiodine whole body scan, computed tomography [CT], magnetic resonance imaging [MRI], or positron emission tomography [PET])
Disease recurrence after 3, 5 and 10 years from the primary treatment | 3, 5 and 10 years from the primary treatment
  Rate of disease recurrence after 3, 5 and 10 years from the primary treatment, detected by any of the available imaging tools (neck sonography, radioiodine whole body scan, computed tomography [CT], magnetic resonance imaging [MRI], or positron emission tomography [PET])
Response to primary therapy | 1, 3, 5 and 10 years after therapy
  Response to primary treatment, evaluated according to the American Thyroid Association guidelines response to treatment: excellent response, biochemical incomplete response, indeterminate response, or structural incomplete response (combination of serum tumor markers and imaging tools, such as neck sonography, radioiodine whole body scan, computed tomography [CT], magnetic resonance imaging [MRI], or positron emission tomography [PET])
Response to secondary treatments | 1, 3, 5 and 10 years after therapy
  Response to secondary treatments, evaluated according to the American Thyroid Association guidelines response to treatment: excellent response, biochemical incomplete response, indeterminate response, or structural incomplete response (combination of serum tumor markers and imaging tools, such as neck sonography, radioiodine whole body scan, computed tomography [CT], magnetic resonance imaging [MRI], or positron emission tomography [PET])

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiano Filetti, MD, Principal Investigator — Full professor of Internal Medicine
Locations (35):
- Italy (35):
  - A.S.S.T. Grande Ospedale Metropolitano Niguarda, Milan, Milano
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Milano
  - IRCCS Ospedale San Raffaele, Milan, Milano
  - Ospedale Regina Apostolorum, Albano Laziale, RM
  - Ospedali Riuniti di Ancona, Ancona
  - Università degli Studi di Bari, Bari
  - Ospedale degli Infermi di Biella, Biella
  - Azienda Unità Sanitaria di Bologna - Ospedale Maggiore, Bologna
  - University of Bologna, S. Orsola Malpighi Hospital, Bologna
  - Università degli Studi di Brescia, Spedali Civili, Brescia
  - Azienda Ospedaliero-Universitaria di Cagliari, Cagliari
  - Azienda Ospedaliero Universitaria "Mater Domini" di Catanzaro, Catanzaro
  - Azienda Ospedaliero Universitaria di Ferrara, Ferrara
  - University of Florence, Florence
  - Ente Ospedaliero Ospedali Galliera, Genova
  - Sapienza University of Rome, Santa Maria Goretti Hospital, Latina
  - Tinchi Pisticci Hospital, Matera
  - Azienda Ospedaliera Universitaria "Gaetano Martino", Messina
  - Università degli Studi di Milano, Istituto Auxologico, Milan
  - University of Modena and Reggio Emilia, Modena
  - University of Naples Federico II, Napoli
  - Azienda Ospedale-Università Padova, Padua
  - Istituto Oncologico del Veneto IRCCS, Padua
  - University of Parma, Parma
  - Istituti Clinici Scientifici Maugeri, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Bio-Medical Campus University, Roma
  - IRCCS Istituti Fisioterapici Ospitalieri - IFO - Istituto Regina Elena, Roma
  - Sapienza University of Rome, Sant'Andrea Hospital, Roma
  - Sapienza University of Rome, Rome
  - A.O.U. Ruggi d'Aragona, Salerno
  - University of Siena, Siena
  - AOU Città della Salute e della Scienza, Torino
  - University of Turin, Gradenigo Hospital, Torino
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lamartina L, Grani G, Arvat E, Nervo A, Zatelli MC, Rossi R, Puxeddu E, Morelli S, Torlontano M, Massa M, Bellantone R, Pontecorvi A, Montesano T, Pagano L, Daniele L, Fugazzola L, Ceresini G, Bruno R, Rossetto R, Tumino S, Centanni M, Meringolo D, Castagna MG, Salvatore D, Nicolucci A, Lucisano G, Filetti S, Durante C. 8th edition of the AJCC/TNM staging system of thyroid cancer: what to expect (ITCO#2). Endocr Relat Cancer. 2018 Mar;25(3):L7-L11. doi: 10.1530/ERC-17-0453. Epub 2017 Nov 30. No abstract available. PMID 29192093
- [Result] Lamartina L, Durante C, Lucisano G, Grani G, Bellantone R, Lombardi CP, Pontecorvi A, Arvat E, Felicetti F, Zatelli MC, Rossi R, Puxeddu E, Morelli S, Torlontano M, Crocetti U, Montesano T, Giubbini R, Orlandi F, Aimaretti G, Monzani F, Attard M, Francese C, Antonelli A, Limone P, Rossetto R, Fugazzola L, Meringolo D, Bruno R, Tumino S, Ceresini G, Centanni M, Monti S, Salvatore D, Spiazzi G, Mian C, Persani L, Barbaro D, Nicolucci A, Filetti S. Are Evidence-Based Guidelines Reflected in Clinical Practice? An Analysis of Prospectively Collected Data of the Italian Thyroid Cancer Observatory. Thyroid. 2017 Dec;27(12):1490-1497. doi: 10.1089/thy.2017.0299. Epub 2017 Nov 10. PMID 29020892
- [Result] Grani G, Zatelli MC, Alfo M, Montesano T, Torlontano M, Morelli S, Deandrea M, Antonelli A, Francese C, Ceresini G, Orlandi F, Maniglia CA, Bruno R, Monti S, Santaguida MG, Repaci A, Tallini G, Fugazzola L, Monzani F, Giubbini R, Rossetto R, Mian C, Crescenzi A, Tumino D, Pagano L, Pezzullo L, Lombardi CP, Arvat E, Petrone L, Castagna MG, Spiazzi G, Salvatore D, Meringolo D, Solaroli E, Monari F, Magri F, Triggiani V, Castello R, Piazza C, Rossi R, Ferraro Petrillo U, Filetti S, Durante C. Real-World Performance of the American Thyroid Association Risk Estimates in Predicting 1-Year Differentiated Thyroid Cancer Outcomes: A Prospective Multicenter Study of 2000 Patients. Thyroid. 2021 Feb;31(2):264-271. doi: 10.1089/thy.2020.0272. Epub 2020 Jul 1. PMID 32475305
- [Result] Forleo R, Grani G, Alfo M, Zilioli V, Giubbini R, Zatelli MC, Gagliardi I, Piovesan A, Ragni A, Morelli S, Puxeddu E, Pagano L, Deandrea M, Ceresini G, Torlontano M, Puligheddu B, Antonelli A, Centanni M, Fugazzola L, Spiazzi G, Monti S, Rossetto R, Monzani F, Tallini G, Crescenzi A, Sparano C, Bruno R, Repaci A, Tumino D, Pezzullo L, Lombardi CP, Ferraro Petrillo U, Filetti S, Durante C, Castagna MG. Minimal Extrathyroidal Extension in Predicting 1-Year Outcomes: A Longitudinal Multicenter Study of Low-to-Intermediate-Risk Papillary Thyroid Carcinoma (ITCO#4). Thyroid. 2021 Dec;31(12):1814-1821. doi: 10.1089/thy.2021.0248. Epub 2021 Oct 20. PMID 34541894
- [Result] Grani G, Gentili M, Siciliano F, Albano D, Zilioli V, Morelli S, Puxeddu E, Zatelli MC, Gagliardi I, Piovesan A, Nervo A, Crocetti U, Massa M, Sama MT, Mele C, Deandrea M, Fugazzola L, Puligheddu B, Antonelli A, Rossetto R, D'Amore A, Ceresini G, Castello R, Solaroli E, Centanni M, Monti S, Magri F, Bruno R, Sparano C, Pezzullo L, Crescenzi A, Mian C, Tumino D, Repaci A, Castagna MG, Triggiani V, Porcelli T, Meringolo D, Locati L, Spiazzi G, Di Dalmazi G, Anagnostopoulos A, Leonardi S, Filetti S, Durante C. A Data-Driven Approach to Refine Predictions of Differentiated Thyroid Cancer Outcomes: A Prospective Multicenter Study. J Clin Endocrinol Metab. 2023 Jul 14;108(8):1921-1928. doi: 10.1210/clinem/dgad075. PMID 36795619
- See also: ITCO Foundation homepage — http://www.itcofoundation.org